CLINICAL TRIAL: NCT05732831
Title: A Phase 1/2, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, and Preliminary Anti-tumor Activity of TNG462 as a Single Agent and in Combination in Patients With MTAP-deleted Advanced or Metastatic Solid Tumors
Brief Title: Safety and Tolerability of TNG462 in Patients With MTAP-deleted Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tango Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG462-C101
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Solid Tumor
Keywords: MTAP deletion; PRMT5; cholangiocarcinoma; NSCLC; mesothelioma; MPNST; Tango; pancreatic; sarcoma; urothelial; gallbladder; liver; renal; breast
MeSH Terms: conditions — Cholangiocarcinoma; Mesothelioma; Neurofibrosarcoma; Sarcoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation (sequential) followed by phase 2 dose expansion in 5 arms (parallel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation (Experimental): Participants with MTAP-deleted solid tumors (excluding primary CNS) will receive escalating doses of TNG462 single agent and in combination with pembrolizumab to estimate the MTD
  Interventions: Drug: TNG462; Drug: Pembrolizumab
- Dose Expansion in NSCLC (Experimental): Participants with MTAP-deleted NSCLC (squamous and non squamous) will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462
- Dose Expansion in Mesothelioma (Experimental): Participants with MTAP-deleted mesothelioma will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462
- Dose Expansion in Pancreatic Ductal Adenocarcinoma (Experimental): Participants with MTAP-deleted pancreatic ductal adenocarcinoma will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462
- Dose Expansion in Sarcoma (Experimental): Participants with MTAP-deleted sarcoma (soft tissue or bone) will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462
- Dose Expansion in Solid Tumors (Experimental): Participants with other MTAP-deleted solid tumors will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462
- Dose Expansion in NSCLC in Combination with Pembrolizumab (Experimental): Participants NSCLC (squamous and non squamous) MTAP-deleted solid tumors will receive TNG462 at the identified RP2D(s)
  Interventions: Drug: TNG462; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TNG462 — TNG462, a selective PRMT5 inhibitor, will be administered orally
Drug: Pembrolizumab — An anti PD-1 antibody, will be administered intravenously
  Other Names: Keytruda
  Arms: Dose Escalation; Dose Expansion in NSCLC in Combination with Pembrolizumab

SUMMARY:
This is a first in human study in patients with advanced or metastatic solid tumors known to have an MTAP deletion. The first part of the study is an open-label, dose escalation and the second part is an open label dose expansion in specific MTAP-deleted tumor types. The study drug, TNG462, is a selective PRMT5 inhibitor administered orally. The study is planned to treat up to 225 participants.

DETAILED DESCRIPTION:
This is a Phase 1/2 multi-center, open label study in solid tumor patients who have a confirmed homozygous MTAP deletion in their tumor. The Phase 1 portion is a dose escalation study of oral TNG462 administered as a single agent and in combination with pembrolizumab in patients with confirmed MTAP-deleted solid tumors. In Phase 2, 6 expansion arms defined by confirmed MTAP-deleted tumor types will enroll in parallel at the RP2D(s) of TNG462 and in combination. In both parts of the study participants who tolerate the drug may continue treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years-of-age at the time of signature of the main study ICF
2. Performance status: ECOG Performance Score of 0 to 1
3. Confirmed histologic or cytologic diagnosis of a locally advanced, metastatic, and/or unresectable solid tumor
4. Prior standard therapy, as available
5. Documented bi-allelic (homozygous) deletion of MTAP in a tumor detected by next- generation sequencing or absence of MTAP protein in a tumor detected by IHC.
6. Adequate organ function/reserve per local labs
7. Adequate liver function per local labs
8. Adequate renal function per local labs
9. Negative serum pregnancy test result at screening
10. Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to TNG462, or its excipients or to pembrolizumab in the combination treatment arms
2. Uncontrolled intercurrent illness that will limit compliance with the study requirements
3. Active infection requiring systemic therapy
4. Currently participating in or has planned participation in a study of another investigational agent or device
5. Impairment of GI function or disease that may significantly alter the absorption of oral TNG462
6. Active prior or concurrent malignancy.
7. Central nervous system metastases associated with progressive neurological symptoms
8. Current active liver disease from any cause
9. Known to be HIV positive, unless all of the following criteria are met:

   1. CD4+ count ≥300/μL
   2. Undetectable viral load
   3. Receiving highly active antiretroviral therapy
10. Clinically relevant cardiovascular disease
11. A female patient who is pregnant or lactating
12. Patient is unwilling or unable to comply with the scheduled visits, drug administration plan, laboratory tests, biopsy, or other study procedures and study restrictions
13. Patient has a prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, may affect the safety of the patient or impair the assessment of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Maximum Tolerated Dose | 28 days and 21 days
  To determine the maximum tolerated dose (MTD) of TNG462 when administered as a single agent and in combination with pembrolizumab
Phase 1 Dosing Schedule | 28 days
  To determine the dosing schedule of TNG462
Phase 2 Anti-neoplastic Activity | 16 weeks and 18 weeks
  To assess anti-neoplastic activity of TNG462 administered single agent and in combination with pembrolizumab in patients with MTAP-deleted advanced solid tumors by RECIST v1.1, iRECIST or mRECIST v1.1

SECONDARY OUTCOMES:
Phase 1 Anti-neoplastic Activity | 16 weeks
  To assess preliminary evidence of anti-neoplastic activity of TNG462 as a single agent and when administered in combination with pembrolizumab in patients with MTAP-deleted advanced solid tumors by RECIST v1.1, iRECIST or mRECIST v1.1
Phase 1 and 2 Adverse Event Profile | 28 days and 21 days
  To describe the safety and tolerability profile of TNG462 by frequency and severity of AEs
Phase 1 and 2 Concentration versus Time Curve | 16 days
  Measure the area under the plasma concentration versus time curve (AUC)
Phase 1 and 2 Time to Achieve Maximal Plasma Concentration | 16 days
  Measure the time to achieve maximal plasma concentration (Tmax)
Phase 1 and 2 Maximum Observed Plasma Concentration | 16 days
  Measure the maximum observed plasma concentration (Cmax)
Phase 1 and 2 Terminal Elimination Half-life | 16 days
  Determine the terminal elimination half-life (t1/2)
Phase 1 and 2 Total Plasma Clearance | 16 days
  Determine the apparent total plasma clearance when dosed orally (CL/F)
Phase 1 and 2 Volume of Distribution | 16 days
  Determine the apparent volume of distribution when dosed orally (Vz/F)
Phase 1 and 2 SDMA Levels | 28 days
  SDMA levels in tumor tissue will be assessed pre-treatment and post treatment with TNG462

CONTACTS AND LOCATIONS:
Overall Officials: Maeve Waldron-Lynch, MD, Study Director — Tango Therapeutics, Inc.
Locations (26):
- United States (15):
  - Stanford University, Palo Alto, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University Chicago Medicine, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Midwestern Regional Medical Center, City of Hope Chicago, Zion, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Center, Detroit, Michigan
  - New York University Langone Health, New York, New York
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Next Oncology Virginia, Fairfax, Virginia
- France (4):
  - CHU de Brest, Brest
  - Centre Berard Leon, Lyon
  - Institut de Cancerologie de l'Ouest - Hôpital Saint Herblain - PPDS, Saint-Herblain
  - Institute Gustav Roussy, Villejuif
- Spain (7):
  - Vall d'Hebron Barcelona Hospital, Barcelona, Catalonia
  - Hospital HM Nou Delfos, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital de Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No